CLINICAL TRIAL: NCT05391828
Title: Randomized Control Trial Comparing Zimmer Biomet Persona Medial Congruent Versus Posterior Stabilized Total Knee Arthroplasty for Treatment of Knee Arthritis Using the ROSA Knee System
Brief Title: Persona MC vs PS RCT With ROSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-00033
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Total Knee Arthroplasty (TKA) performed using a medial congruent articular bearing surface design (Experimental)
  Interventions: Device: Zimmer-Biomet Persona Medial Congruent (MC) Bearing Design
- Total Knee Arthroplasty (TKA) performed using a posterior stabilized bearing design (Active Comparator)
  Interventions: Device: Zimmer-Biomet Persona Posterior-Stabilized (PS) Bearing Design

INTERVENTIONS:
Device: Zimmer-Biomet Persona Medial Congruent (MC) Bearing Design — TKA will be performed using the MC Bearing Design. The MC bearing provides medial stability and lateral mobility to facilitate more natural motion.
  Arms: Total Knee Arthroplasty (TKA) performed using a medial congruent articular bearing surface design
Device: Zimmer-Biomet Persona Posterior-Stabilized (PS) Bearing Design — TKA will be performed using the PS Bearing Design. The PS bearings are designed to provide ±1.5 degrees varus/valgus constraint and ± 5.5 degrees internal/external rotation constraint.
  Arms: Total Knee Arthroplasty (TKA) performed using a posterior stabilized bearing design

SUMMARY:
A randomized, controlled study comparing two total knee implant devices, Persona medial congruent (MC) vs posterior stabilized (PS). These surgeries will be performed using the ROSA robotic system. Patients will be followed up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years of age
2. Patients scheduled an elective primary TKA for a diagnosis of osteoarthritis or inflammatory arthritis using the ROSA Knee System.
3. Patient is willing to cooperate and follow study protocol and visit schedule
4. Subject has access to a device is capable of pairing to the Apple Watch, supporting application updates and is compatible with the mymobility App.

Exclusion Criteria:

1. Patient is pregnant
2. Patient is unable to provide written consent
3. Revision TKA
4. History of prior infection in the affected knee
5. History of prior open surgery with significant hardware in place on the affected knee (i.e. prior distal femur or proximal tibia fracture or osteotomy)
6. Preoperative diagnosis of post-traumatic arthritis, avascular necrosis, or fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR) | Baseline
  KOOS, JR contains 7 items from the original KOOS survey. Items are coded from 0 to 4, none to extreme respectively. KOOS, JR is scored by summing the raw response (range 0-28) and then converting it to an interval score. The interval score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR) | Week 6
  KOOS, JR contains 7 items from the original KOOS survey. Items are coded from 0 to 4, none to extreme respectively. KOOS, JR is scored by summing the raw response (range 0-28) and then converting it to an interval score. The interval score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR) | Month 3
  KOOS, JR contains 7 items from the original KOOS survey. Items are coded from 0 to 4, none to extreme respectively. KOOS, JR is scored by summing the raw response (range 0-28) and then converting it to an interval score. The interval score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR) | Year 1
  KOOS, JR contains 7 items from the original KOOS survey. Items are coded from 0 to 4, none to extreme respectively. KOOS, JR is scored by summing the raw response (range 0-28) and then converting it to an interval score. The interval score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR) | Year 2
  KOOS, JR contains 7 items from the original KOOS survey. Items are coded from 0 to 4, none to extreme respectively. KOOS, JR is scored by summing the raw response (range 0-28) and then converting it to an interval score. The interval score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR) | Year 5
  KOOS, JR contains 7 items from the original KOOS survey. Items are coded from 0 to 4, none to extreme respectively. KOOS, JR is scored by summing the raw response (range 0-28) and then converting it to an interval score. The interval score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR) | Year 10
  KOOS, JR contains 7 items from the original KOOS survey. Items are coded from 0 to 4, none to extreme respectively. KOOS, JR is scored by summing the raw response (range 0-28) and then converting it to an interval score. The interval score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR) | Year 20
  KOOS, JR contains 7 items from the original KOOS survey. Items are coded from 0 to 4, none to extreme respectively. KOOS, JR is scored by summing the raw response (range 0-28) and then converting it to an interval score. The interval score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.
Forgotten Joint Score (FJS) | Baseline
  FJS is a patient-reported outcome measure intended to determine a patient's ability to "forget" about their affected joint after surgery or treatment. FJS consists of 12 questions - the total score range is 0-100. The higher the score, the less the patient is aware of their affected joint when performing daily activities.
Forgotten Joint Score (FJS) | Week 6
  FJS is a patient-reported outcome measure intended to determine a patient's ability to "forget" about their affected joint after surgery or treatment. FJS consists of 12 questions - the total score range is 0-100. The higher the score, the less the patient is aware of their affected joint when performing daily activities.
Forgotten Joint Score (FJS) | Month 3
  FJS is a patient-reported outcome measure intended to determine a patient's ability to "forget" about their affected joint after surgery or treatment. FJS consists of 12 questions - the total score range is 0-100. The higher the score, the less the patient is aware of their affected joint when performing daily activities.
Forgotten Joint Score (FJS) | Year 1
  FJS is a patient-reported outcome measure intended to determine a patient's ability to "forget" about their affected joint after surgery or treatment. FJS consists of 12 questions - the total score range is 0-100. The higher the score, the less the patient is aware of their affected joint when performing daily activities.
Forgotten Joint Score (FJS) | Year 2
  FJS is a patient-reported outcome measure intended to determine a patient's ability to "forget" about their affected joint after surgery or treatment. FJS consists of 12 questions - the total score range is 0-100. The higher the score, the less the patient is aware of their affected joint when performing daily activities.
Forgotten Joint Score (FJS) | Year 5
  FJS is a patient-reported outcome measure intended to determine a patient's ability to "forget" about their affected joint after surgery or treatment. FJS consists of 12 questions - the total score range is 0-100. The higher the score, the less the patient is aware of their affected joint when performing daily activities.
Forgotten Joint Score (FJS) | Year 10
  FJS is a patient-reported outcome measure intended to determine a patient's ability to "forget" about their affected joint after surgery or treatment. FJS consists of 12 questions - the total score range is 0-100. The higher the score, the less the patient is aware of their affected joint when performing daily activities.
Forgotten Joint Score (FJS) | Year 20
  FJS is a patient-reported outcome measure intended to determine a patient's ability to "forget" about their affected joint after surgery or treatment. FJS consists of 12 questions - the total score range is 0-100. The higher the score, the less the patient is aware of their affected joint when performing daily activities.
European Quality of Life Five Dimension (EQ-5D) Score | Baseline
  The EQ-5D comprises five questions on mobility, self care, pain, usual activities, and psychological status with three possible answers for each item (1=no problem, 2=moderate problem, 3=severe problem. A summary index with a maximum score of 1 can be derived from these five dimensions by conversion with a table of scores. The maximum score of 1 indicates the best health state, by contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems. In addition, there is a visual analogue scale (VAS) to indicate the general health status (0-100) with 100 indicating the best health status.
European Quality of Life Five Dimension (EQ-5D) Score | Week 6
  The EQ-5D comprises five questions on mobility, self care, pain, usual activities, and psychological status with three possible answers for each item (1=no problem, 2=moderate problem, 3=severe problem. A summary index with a maximum score of 1 can be derived from these five dimensions by conversion with a table of scores. The maximum score of 1 indicates the best health state, by contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems. In addition, there is a visual analogue scale (VAS) to indicate the general health status (0-100) with 100 indicating the best health status.
European Quality of Life Five Dimension (EQ-5D) Score | Month 3
  The EQ-5D comprises five questions on mobility, self care, pain, usual activities, and psychological status with three possible answers for each item (1=no problem, 2=moderate problem, 3=severe problem. A summary index with a maximum score of 1 can be derived from these five dimensions by conversion with a table of scores. The maximum score of 1 indicates the best health state, by contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems. In addition, there is a visual analogue scale (VAS) to indicate the general health status (0-100) with 100 indicating the best health status.
European Quality of Life Five Dimension (EQ-5D) Score | Year 1
  The EQ-5D comprises five questions on mobility, self care, pain, usual activities, and psychological status with three possible answers for each item (1=no problem, 2=moderate problem, 3=severe problem. A summary index with a maximum score of 1 can be derived from these five dimensions by conversion with a table of scores. The maximum score of 1 indicates the best health state, by contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems. In addition, there is a visual analogue scale (VAS) to indicate the general health status (0-100) with 100 indicating the best health status.
European Quality of Life Five Dimension (EQ-5D) Score | Year 2
  The EQ-5D comprises five questions on mobility, self care, pain, usual activities, and psychological status with three possible answers for each item (1=no problem, 2=moderate problem, 3=severe problem. A summary index with a maximum score of 1 can be derived from these five dimensions by conversion with a table of scores. The maximum score of 1 indicates the best health state, by contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems. In addition, there is a visual analogue scale (VAS) to indicate the general health status (0-100) with 100 indicating the best health status.
European Quality of Life Five Dimension (EQ-5D) Score | Year 5
  The EQ-5D comprises five questions on mobility, self care, pain, usual activities, and psychological status with three possible answers for each item (1=no problem, 2=moderate problem, 3=severe problem. A summary index with a maximum score of 1 can be derived from these five dimensions by conversion with a table of scores. The maximum score of 1 indicates the best health state, by contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems. In addition, there is a visual analogue scale (VAS) to indicate the general health status (0-100) with 100 indicating the best health status.
European Quality of Life Five Dimension (EQ-5D) Score | Year 10
  The EQ-5D comprises five questions on mobility, self care, pain, usual activities, and psychological status with three possible answers for each item (1=no problem, 2=moderate problem, 3=severe problem. A summary index with a maximum score of 1 can be derived from these five dimensions by conversion with a table of scores. The maximum score of 1 indicates the best health state, by contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems. In addition, there is a visual analogue scale (VAS) to indicate the general health status (0-100) with 100 indicating the best health status.
European Quality of Life Five Dimension (EQ-5D) Score | Year 20
  The EQ-5D comprises five questions on mobility, self care, pain, usual activities, and psychological status with three possible answers for each item (1=no problem, 2=moderate problem, 3=severe problem. A summary index with a maximum score of 1 can be derived from these five dimensions by conversion with a table of scores. The maximum score of 1 indicates the best health state, by contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems. In addition, there is a visual analogue scale (VAS) to indicate the general health status (0-100) with 100 indicating the best health status.

SECONDARY OUTCOMES:
Change in Average gait speed | Baseline, Year 2
Change in Average daily step count | Baseline, Year 2
Change in Average daily flight count | Baseline, Year 2

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Aggarwal, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to Vinay.Aggarwal@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.